CLINICAL TRIAL: NCT05543616
Title: A MASTER PHASE 1/2/3 PROTOCOL TO INVESTIGATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF VARIANT-ADAPTED BNT162b2 RNA-BASED VACCINE CANDIDATE(S) IN HEALTHY CHILDREN
Brief Title: A Study to Learn About Variant-Adapted COVID-19 RNA Vaccine Candidate(s) in Healthy Children
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C4591048; 2024-000001-33 (EudraCT Number); 2023-503736-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Virus; Severe Acute Respiratory Syndrome Coronavirus 2; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (23):
- 3 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 3 microgram dose
- 6 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 6 microgram dose
- 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 1) - 0/8 week schedule (Experimental): Injection in the muscle at 0- and 8-weeks
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 2) - 0/8 week schedule (Experimental): Injection in the muscle at 0- and 8-weeks
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 3 microgram dose, 6 Months to <4 Years 6 Months (Substudy B, Group 1) (Experimental): Injection in the muscle, 2 doses 2 months apart
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose
- 3 microgram dose, 6 Months to <5 Years (Substudy B, Group 2) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose
- 3 microgram dose, 6 Months to <5 Years (Substudy B, Group 3) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose
- 6 microgram dose, 6 Months to <2 Years (Substudy C, Phase 1) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose
- 10 microgram dose, 6 Months to <2 Years (Substudy C, Phase 1) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 10 microgram dose, 5 to <12 Years (Substudy D, Group 1) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 10 microgram dose, 5 to <12 Years (Substudy D, Group 2) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 10 microgram dose, 5 to <12 Years (Substudy D, Group 3) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 3 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 3 microgram dose
- 6 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 6 microgram dose; Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1) (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks and approximately 6-months post-Dose 3
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 6 microgram dose, 2 Years to <5 Years (Substudy C, Phase 1) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose
- 10 microgram dose, 2 Years to <5 Years (Substudy C, Phase 1) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- 3 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 3) - 0/3/11 week schedule (Experimental): Injection in the muscle at 0-, 3-, and 11-weeks
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 3 microgram dose
- 10 microgram dose, 2 to <5 Years (Substudy A, Phase 2/3, Group 4) - Single dose (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 2 to <5 Years (Substudy A, Phase 2/3, Group 5) - Single dose (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 5 Years to <12 Years (Substudy E, Group 2) (Experimental): Injection in the muscle, 1 dose
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose
- 10 microgram dose, 6 months to <2 years (Substudy A Phase 2/3, Group 6) - 0/8 week schedule (Experimental): Injection in the muscle at 0- and 8-weeks
  Interventions: Biological: Variant-adapted BNT162b2 (Omicron KP.2) 10 microgram dose

INTERVENTIONS:
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose — Injection in the muscle
  Arms: 3 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1); 3 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1); 3 microgram dose, 6 Months to <4 Years 6 Months (Substudy B, Group 1); 3 microgram dose, 6 Months to <5 Years (Substudy B, Group 2); 3 microgram dose, 6 Months to <5 Years (Substudy B, Group 3)
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose — Injection in the muscle
  Arms: 6 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1); 6 microgram dose, 2 Years to <5 Years (Substudy C, Phase 1); 6 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1); 6 microgram dose, 6 Months to <2 Years (Substudy C, Phase 1)
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose — Injection in the muscle
  Arms: 10 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1); 10 microgram dose, 2 Years to <5 Years (Substudy C, Phase 1); 10 microgram dose, 5 to <12 Years (Substudy D, Group 1); 10 microgram dose, 5 to <12 Years (Substudy D, Group 2); 10 microgram dose, 5 to <12 Years (Substudy D, Group 3); 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1); 10 microgram dose, 6 Months to <2 Years (Substudy C, Phase 1)
Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 3 microgram dose — Injection in the muscle
  Arms: 3 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1); 3 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1); 3 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 3) - 0/3/11 week schedule
Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 6 microgram dose — Injection in the muscle
  Arms: 6 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1); 6 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1)
Biological: Variant-adapted BNT162b2 (Omicron XBB.1.5) 10 microgram dose — injection in the muscle
  Arms: 10 microgram dose, 2 to <5 Years (Substudy A, Phase 2/3, Group 4) - Single dose; 10 microgram dose, 2 to <5 Years (Substudy A, Phase 2/3, Group 5) - Single dose; 10 microgram dose, 5 Years to <12 Years (Substudy E, Group 2); 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 1); 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 1) - 0/8 week schedule; 10 microgram dose, 6 Months to <2 Years (Substudy A, Phase 2/3, Group 2) - 0/8 week schedule; 6 microgram dose, 2 Years to <4 years 3 months (Substudy A, Phase 1)
Biological: Variant-adapted BNT162b2 (Omicron KP.2) 10 microgram dose — Injection in the muscle
  Arms: 10 microgram dose, 6 months to <2 years (Substudy A Phase 2/3, Group 6) - 0/8 week schedule

SUMMARY:
The purpose of this clinical trial is to learn about the safety, extent of the side effects, and immune responses of the study vaccine (called variant-adapted BNT162b2 RNA-based vaccine) in healthy children. The trial is divided into 5 individual studies or substudies based on age group and prior history of COVID-19 vaccinations. All participants in each of the 5 sub-studies will receive study vaccine as a shot depending on what group they are in.

* Substudy A design: Phase 1 includes participants 6 months through less than 4 years 3 months of age who have not received a previous coronavirus vaccination (COVID-19 vaccine naïve) and will receive 3 doses of study vaccine as their initial series, followed by a fourth dose of study vaccine. Phase 2/3 includes participants 6 months through less than 5 years of age who have not received a previous coronavirus vaccination (COVID-19 vaccine naive) and will receive 1, 2, or 3 doses of study vaccine, depending on what group they are in.
* Substudy B design: includes participants 6 months through less than 5 years of age who have either received 2 or 3 prior doses of BNT162b2 and will receive study vaccine as their third or fourth dose.
* Substudy C design: Phase 1 includes participants 6 months through less than 5 years of age who have received 3 prior doses of BNT162b2 and will receive study vaccine as their fourth dose.
* Substudy D design: includes participants 5 through less than12 years of age who have received 2 or 3 prior doses of BNT162b2 and will receive study vaccine as their third or fourth dose.
* Substudy E design: includes participants 5 through less than 12 years of age who have not received a previous coronavirus vaccination (COVID-19 vaccine naive) and will receive a single dose of study vaccine.

ELIGIBILITY:
Substudy A

Inclusion Criteria:

* Phase 1: Healthy male or female participants ≥6 months to <4 years 3 months of age, at the time of randomization.
* Phase 2/3: Healthy male or female participants ≥6 months to <5 years of age at the time of randomization/enrollment.

Exclusion Criteria:

* Previous or current diagnosis of multisystem inflammatory syndrome in children (MIS-C).
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, or individuals who receive treatment with immunosuppressive therapy.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus. Note: Stable type 1 diabetes and hypothyroidism are permitted.
* Any history of myocarditis or pericarditis.
* Previous vaccination with any COVID-19 vaccine.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer) or radiotherapy, within 60 days before enrollment through the conclusion of the study. Systemic corticosteroids (≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) for ≥14 days is prohibited from 28 days prior to enrollment through 28 days after administration of study intervention.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.

Substudy B

Inclusion Criteria:

- Healthy male or female participants = ≥6 months to <5 years of age, at the time of enrollment.

Exclusion Criteria:

* Previous or current diagnosis of MIS-C.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, or individuals who receive treatment with immunosuppressive therapy.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus.
* Prior receipt of any COVID 19 vaccine other than BNT162b2.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer) or radiotherapy, within 60 days before enrollment through the conclusion of the study. Systemic corticosteroids (≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) for ≥14 days is prohibited from 28 days prior to enrollment through 28 days after administration of study intervention.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.

Substudy C

Inclusion Criteria:

- Healthy male or female participants ≥6 months to <5 years of age, at the time of randomization/enrollment.

Exclusion Criteria:

* Previous or current diagnosis of MIS-C.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, or individuals who receive treatment with immunosuppressive therapy.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus.
* Prior receipt of any COVID 19 vaccine other than BNT162b2.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer) or radiotherapy, within 60 days before enrollment through the conclusion of the study. Systemic corticosteroids (≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) for ≥14 days is prohibited from 28 days prior to enrollment through 28 days after administration of study intervention.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.

Substudy D

Inclusion Criteria:

- Healthy male or female participants ≥5 years to <12 years of age, at the time of enrollment.

Exclusion Criteria:

* Previous or current diagnosis of MIS-C.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, or individuals who receive treatment with immunosuppressive therapy.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus.
* Female who is pregnant or breastfeeding.
* Prior receipt of any COVID 19 vaccine other than BNT162b2.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer) or radiotherapy, within 60 days before enrollment through the conclusion of the study. Systemic corticosteroids (≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) for ≥14 days is prohibited from 28 days prior to enrollment through 28 days after administration of study intervention.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.

Substudy E

Inclusion Criteria:

- Healthy male or female participants ≥5 years to <12 years of age, at the time of enrollment.

Exclusion Criteria:

* Previous or current diagnosis of MIS-C.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination, or individuals who receive treatment with immunosuppressive therapy.
* Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus.
* Any history of myocarditis or pericarditis.
* Female who is pregnant or breastfeeding.
* Previous vaccination with any COVID 19 vaccine.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer) or radiotherapy, within 60 days before enrollment through the conclusion of the study. Systemic corticosteroids (≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) for ≥14 days is prohibited from 28 days prior to enrollment through 28 days after administration of study intervention.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4292 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Substudy A (SSA) - Ph 1 dose finding, percentage of participants reporting local reactions | for up to 7 days following Dose 1, Dose 2, Dose 3 and Dose 4
  Participants ≥6 months to <2 years of age: tenderness at the injection site, redness, and swelling as self-reported on electronic diaries Participants ≥2 to <5 years of age: pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSA - Ph 1 dose finding, percentage of participants reporting systemic events | for up to 7 days following Dose 1, Dose 2, Dose 3 and Dose 4
  Participants ≥6 months to <2 years of age: fever, decreased appetite, drowsiness, and irritability as self-reported on electronic diaries Participants ≥2 to <5 years of age: fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSA - Ph 1 dose finding, percentage of participants reporting adverse events | from Dose 1 to 1 month after Dose 3 and from Dose 4 to 1 month after Dose 4
  as elicited by investigational site staff
SSA - Ph 1 dose finding, percentage of participants reporting serious adverse events | from Dose 1 to 6 months after the last dose
  as elicited by investigational site staff
SSA - Ph 2/3, percentage of participants reporting local reactions | for up to 7 days following Dose 1 (for Groups 1 through 6), Dose 2 (for Groups 1, 2, 3, and 6), and Dose 3 (for Group 3)
  Participants ≥6 months to <2 years of age: tenderness at the injection site, redness, and swelling as self-reported on electronic diaries Participants ≥2 to <5 years of age: pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSA - Ph 2/3, percentage of participants reporting systemic events | for up to 7 days following Dose 1 (for Groups 1 through 6), Dose 2 (for Groups 1, 2, 3, and 6), and Dose 3 (for Group 3)
  Participants ≥6 months to <2 years of age: fever, decreased appetite, drowsiness, and irritability as self-reported on electronic diaries Participants ≥2 to <5 years of age: fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSA - Ph 2/3, percentage of participants reporting adverse events | from Dose 1 to 1 month after the last dose
  as elicited by investigational site staff
SSA - Ph 2/3, percentage of participants reporting serious adverse events | from Dose 1 to 6 months after the last dose
  as elicited by investigational site staff
SSA - Ph 2/3, noninferiority with respect to ratio of the geometric mean of SARS-CoV-2 Omicron XBB.1.5-neutralizing titers in participants ≥6 months to <2 years of age | At 1 month after 2 doses of BNT162b2 (Omicron XBB.1.5) 10 microgram (on a 0- and 8-week schedule) to 1 month after 3 doses (on a 0-, 3-, and 11-week schedule) of BNT162b2 (Omicron XBB.1.5) 3 microgram
  As measured at the central laboratory
SSA - Ph 2/3, noninferiority with respect to seroresponse rate to the Omicron XBB.1.5 strain titers in participants ≥6 months to <2 years of age | At 1 month after 2 doses of BNT162b2 (Omicron XBB.1.5) 10 microgram (on a 0- and 8-week schedule) and at 1 month after 3 doses (on a 0-, 3-, and 11-week schedule) of BNT162b2 (Omicron XBB.1.5) 3 microgram
  As measured at the central laboratory
SSA - Ph 2/3, noninferiority with respect to ratio of the geometric mean of SARS-CoV-2 Omicron XBB.1.5-neutralizing titers in participants ≥2 to <5 years of age | At 1 month after 1 dose of BNT162b2 (Omicron XBB.1.5) 10 microgram in participants ≥2 to <5 years of age to 1 month after 3 doses (on a 0/3/11-week schedule) of BNT162b2 (Omicron XBB.1.5) 3 microgram in participants ≥6 months to <2 years of age
  As measured at the central laboratory
SSA - Ph 2/3, noninferiority with respect to seroresponse rate to the Omicron XBB.1.5 strain in participants ≥2 to <5 years of age | At 1 month after 1 dose of BNT162b2 (Omicron XBB.1.5) 10 microgram in participants ≥2 to <5 years of age and at 1 month after 3 doses (0/3/11-week schedule) of BNT162b2 (Omicron XBB.1.5) 3 microgram in participants ≥6 months to <2 years of age
  As measured at the central laboratory
Substudy B (SSB) - percentage of participants reporting local reactions | for up to 7 days following Dose 1 (for Groups 1, 2 and 3) and Dose 2 (for Group 1)
  Participants ≥6 months to <2 years of age: tenderness at the injection site, redness, and swelling as self-reported on electronic diaries Participants ≥2 to <5 years of age: pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSB - percentage of participants reporting systemic events | for up to 7 days following Dose 1 (for Groups 1, 2 and 3) and Dose 2 (for Group 1)
  Participants ≥6 months to <2 years of age: fever, decreased appetite, drowsiness, and irritability as self-reported on electronic diaries Participants ≥2 to <5 years of age: fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSB - percentage of participants reporting adverse events | from the first study vaccination to 1 month after the first study vaccination (for Groups 1, 2, and 3), and from the second study vaccination to 1 month after the second study vaccination (for Group 1 only)
  as elicited by investigational site staff
SSB - percentage of participants reporting serious adverse events | from Dose 1 to 6 months after the last dose
  as elicited by investigational site staff
SSB - superiority with respect to ratio of the geometric mean of SARS-CoV-2 Omicron BA.4/BA.5-neutralizing titers in participants ≥6 months to <5 years of age | at 1 month after Dose 4 for Group 2 participants who received 3 prior doses of BNT162b2 3 µg and a fourth dose of bivalent BNT162b2 to 1 month after Dose 3 in Study C4591007 participants ≥6 months to <5 years of age who received 3 doses of BNT162b2 3 µg
  As measured at the central laboratory
SSB - noninferiority with respect to seroresponse rate to the Omicron BA.4/BA.5 strain in participants ≥6 months to <5 years of age | at 1 month after Dose 4 for Group 2 participants who received 3 prior doses of BNT162b2 3 µg and a fourth dose of bivalent BNT162b2 to 1 month after Dose 3 in Study C4591007 participants ≥6 months to <5 years of age who received 3 doses of BNT162b2 3 µg
  As measured at the central laboratory
Substudy C (SSC) - Ph 1 dose finding, percentage of participants reporting local reactions | for up to 7 days following Dose 1
  Participants ≥6 months to <2 years of age: tenderness at the injection site, redness, and swelling as self-reported on electronic diaries Participants ≥2 to <5 years of age: pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSC - Ph 1 dose finding, percentage of participants reporting systemic events | for up to 7 days following Dose 1
  Participants ≥6 months to <2 years of age: fever, decreased appetite, drowsiness, and irritability as self-reported on electronic diaries Participants ≥2 to <5 years of age: fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSC - Ph 1 dose finding, percentage of participants reporting adverse events | 1 month after Dose 1
  as elicited by investigational site staff
SSC - Ph 1 dose finding, percentage of participants reporting serious adverse events | 6 months after Dose 1
  as elicited by investigational site staff
SSC - Ph 1 dose finding - geometric mean titers elicited by prophylactic bivalent BNT162b2 at each dose level given as a fourth dose in participants ≥6 months to <5 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSC - Ph 1 dose finding - geometric mean fold rise elicited by prophylactic bivalent BNT162b2 at each dose level given as a fourth dose in participants ≥6 months to <5 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSC - Ph 1 dose finding - percentage of participants with seroresponse elicited by prophylactic bivalent BNT162b2 at each dose level given as a fourth dose in participants ≥6 months to <5 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
Substudy D (SSD) - percentage of participants reporting local reactions | for up to 7 days following Dose 1
  pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSD - percentage of participants reporting systemic events | for up to 7 days following Dose 1
  fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSD - percentage of participants reporting adverse events | 1 month after Dose 1
  as elicited by investigational site staff
SSD - percentage of participants reporting serious adverse events | 6 months after Dose 1
  as elicited by investigational site staff
SSD - the ratio of the geometric mean of SARS-CoV-2 Omicron BA.4/BA.5-neutralizing titers in participants ≥5 to <12 years of age | at 1 month after Dose 4 for participants who received 3 prior doses of BNT162b2 10 μg and a fourth dose of bivalent BNT162b2 to those at 1 month after Dose 3 for Study C4591007 Phase 2/3 participants who received 3 doses of BNT162b2 10 μg
  As measured at the central laboratory
SSD - difference in percentages of participants with seroresponse to the Omicron BA.4/BA.5 strain in participants ≥5 to <12 years of age | at 1 month after bivalent BNT162b2 as a fourth dose for participants who received 3 prior doses of BNT162b2 10 µg and at 1 month after a third dose of BNT162b2 10 µg for Study C4591007 Phase 2/3 participants who received 3 doses of BNT162b2 10 µg
  As measured at the central laboratory
Substudy E (SSE) - percentage of participants reporting local reactions | for up to 7 days following Dose 1
  pain at the injection site, redness, and swelling as self-reported on electronic diaries
SSE - percentage of participants reporting systemic events | for up to 7 days following Dose 1
  fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries
SSE - percentage of participants reporting adverse events | from Dose 1 to 1 month after Dose 1
  as elicited by investigational site staff
SSE - percentage of participants reporting serious adverse events | from Dose 1 to 6 months after Dose 1
  as elicited by investigational site staff
SSE - Ratio of the geometric mean of SARS-CoV-2 Omicron XBB.1.5-neutralizing titers | At 1 month after 1 dose of BNT162b2 (Omi XBB.1.5) 10 microgram in participants ≥5 to 12 years of age to 1 month after 1 dose of BNT162b2 (Omi XBB.1.5) 30 microgram in participants ≥12 years of age from study C4591054 Substudy A
  As measured at the central laboratory
SSE - difference in percentage of participants with seroresponse to Omicron XBB.1.5 | At 1 month after 1 dose of BNT162b2 (Omi XBB.1.5) 10 microgram in participants ≥5 to 12 years of age and 1 month after 1 dose of BNT162b2 (Omi XBB.1.5) 30 microgram in participants ≥12 years of age from study C4591054 Substudy A
  As measured at the central laboratory

SECONDARY OUTCOMES:
SSA - Ph 1 dose finding, geometric mean titers elicited by prophylactic variant-adapted BNT162b2 at each dose level and variant vaccine type (if applicable) in COVID-19 vaccine-naïve participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 2, 1 month after Dose 3, and 1 month after Dose 4
  As measured at the central laboratory
SSA - Ph 1 dose finding, geometric mean fold rise elicited by prophylactic variant-adapted BNT162b2 at each dose level and variant vaccine type (if applicable) in COVID-19 vaccine-naïve participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 2, and 1 month after Dose 3
  As measured at the central laboratory
SSA - Ph 1 dose finding, percentage of participants with seroresponse elicited by prophylactic variant-adapted BNT162b2 at each dose level and variant-adapted vaccine type in COVID-19 vaccine-naïve participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 2, and 1 month after Dose 3
  As measured at the central laboratory
SSA - Ph 2/3, geometric mean titers elicited by variant-adapted BNT162b2 (Omicron XBB.1.5) in COVID-19 vaccine-naive participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 1 (Groups 2 and 4), 1 month after Dose 2 (Group 1), and 1 month after Dose 3 (Group 3)
  As measured at the central laboratory
SSA - Ph 2/3, geometric mean fold rise elicited by variant-adapted BNT162b2 (Omicron XBB.1.5) in COVID-19 vaccine naive participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 1 (Groups 2 and 4), 1 month after Dose 2 (Group 1), and 1 month after Dose 3 (Group 3)
  As measured at the central laboratory
SSA - Ph 2/3, percentages of participants with seroresponse elicited by variant-adapted BNT162b2 (Omicron XBB.1.5) in COVID-19 vaccine-naive participants ≥6 months to <5 years of age | At baseline (before Dose 1), 1 month after Dose 1 (Groups 2 and 4), 1 month after Dose 2 (Group 1), and 1 month after Dose 3 (Group 3)
  As measured at the central laboratory
SSB - geometric mean titers elicited by bivalent BNT162b2 given as third and/or fourth dose in participants ≥6 months <5 years of age | Group 1: At baseline (before Dose 1), 1 month after Dose 1 and 1 month after Dose 2; Groups 2 and 3: At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSB - geometric mean fold rise elicited by bivalent BNT162b2 given as third and/or fourth dose in participants ≥6 months <5 years of age | Group 1: At baseline (before Dose 1), 1 month after Dose 1 and 1 month after Dose 2; Groups 2 and 3: At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSB - percentages of participants with seroresponse elicited by bivalent BNT162b2 given as third and/or fourth dose in participants ≥6 months <5 years of age | Group 1: At baseline (before Dose 1), 1 month after Dose 1 and 1 month after Dose 2; Groups 2 and 3: At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSB - noninferiority with respect to ratio of the geometric mean of SARS-CoV-2 reference strain-neutralizing titers in participants ≥6 months to <5 years of age | at 1 month after Dose 4 for participants who received 3 prior doses of BNT162b2 3 µg and a fourth dose of bivalent BNT162b2 to Study C4591007 participants ≥6 months to <5 years of age who received 3 doses of BNT162b2 3 µg
  As measured at the central laboratory
SSB - noninferiority with respect to seroresponse rate to the reference strain in participants ≥6 months to <5 years of age | at 1 month after Dose 4 for participants who received 3 prior doses of BNT162b2 3 µg and a fourth dose of bivalent BNT162b2 to Study C4591007 participants ≥6 months to <5 years of age who received 3 doses of BNT162b2 3 µg
  As measured at the central laboratory
SSD - geometric mean titers elicited by bivalent BNT162b2 given as a fourth dose in participants ≥5 to <12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSD - geometric mean fold rise elicited by bivalent BNT162b2 given as a fourth dose in participants ≥5 to <12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSD - percentages of participants with seroresponse elicited by bivalent BNT162b2 given as a fourth dose in participants ≥5 to <12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSE - geometric mean titers elicited by BNT162b2 (Omicron XBB.1.5) given as a single 10 microgram dose in participants ≥5 to <12 years of age and as a single 30 microgram dose in Study C4591054 Substudy A participants ≥12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSE - geometric mean fold rise elicited by BNT162b2 (Omicron XBB.1.5) given as a single 10 microgram dose in participants ≥5 to <12 years of age and as a single 30 microgram dose in Study C4591054 Substudy A participants ≥12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory
SSE - percentage of participants with seroresponse elicited by BNT162b2 (Omicron XBB.1.5) given as a single 10 microgram dose in participants ≥5 to <12 years of age and as a single 30 mcg dose in Study C4591054 Substudy A participants ≥12 years of age | At baseline (before Dose 1) and 1 month after Dose 1
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (117):
- United States (93):
  - UAB Child Health Research Unit (CHRU), Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - Advanced Research Center Inc., Anaheim, California
  - Paradigm Clinical Research Centers, Inc, La Mesa, California
  - Hoag Medical Group Foothill Ranch, Lake Forest, California
  - Kaiser Permanente, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Oakland, Oakland, California
  - Clinical and Translational Research Unit (CTRU) & Spectrum Biobank, Palo Alto, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Paradigm Clinical Research, LLC, San Diego, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Stanford University Medical Center, Stanford, California
  - PediaClinic, Highlands Ranch, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale University- Yale Center for Clinical Investigation, New Haven, Connecticut
  - Emerson Clinical Research Institute - Washington - Connecticut Avenue, Washington D.C., District of Columbia
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Meridian Clinical Research, LLC, Washington D.C., District of Columbia
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Accel Research Sites Network- Nona Pediatric Center, Orlando, Florida
  - SEC Clinical Research, Pensacola, Florida
  - Asclepes Research Center - Spring Hill, Spring Hill, Florida
  - PAS Research, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Emory Children's Center Illness Pod, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Emory University Investigational Drug Service, Atlanta, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Saltzer Health, Nampa, Idaho
  - The Iowa Clinic, P.C., Ankeny, Iowa
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Center for Immunization Research Inpatient Unit, Baltimore, Maryland
  - Johns Hopkins Center for Immunization Outpatient Clinic, Baltimore, Maryland
  - Boston medical Center (investigational Pharmacy Services, IP delivery), Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston Medical Center Crosstown Building, Boston, Massachusetts
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Velocity Clinical Research, Hastings, Hastings, Nebraska
  - Velocity Clinical Research, Lincoln, Lincoln, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Meridian Clinical Research, LLC, Binghamton, New York
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Jacobi Medical Center, The Bronx, New York
  - Atrium Health - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Senders Pediatrics, Cleveland, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Coastal Pediatric Research, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cedar Health Research, Dallas, Texas
  - Proactive Clinical Research LLC, Edinburg, Texas
  - Proactive Clinical Research, LLC, Edinburg, Texas
  - ACRC TRIALS / Catalyst Physician Group / Frisco Medical Village, Frisco, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Hospital, Houston, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Dr. Ruben Aleman and Associates, McAllen, Texas
  - ACRC Trials (Administrative Site), Plano, Texas
  - Alliance for Multispecialty Research, LLC, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Seattle Children's- Building Cure, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
- Brazil (8):
  - Obras Sociais Irma Dulce, Salvador, Estado de Bahia
  - Consultoria em Controle de Infecção Hospitalar, Belo Horizonte, Minas Gerais
  - Centro Médico São Francisco, Curitiba, Paraná
  - Centro de Estudos e Pesquisa em Molestias Infecciosas - CPCLIN/RN, Natal, Rio Grande do Norte
  - Hospital de Clínicas de Porto Alegre - Escritório de Projetos e Parcerias Estratégicas, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Puerto Rico (2):
  - Clinical Research Puerto Rico, Guayama
  - University of Puerto Rico - Medical Sciences Campus, San Juan
- South Africa (14):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Jaymed Research, Welkom, Free State
  - REIMED Reiger Park, Boksburg, Gauteng
  - Wits RHI, Johannesburg, Gauteng
  - University of Witwatersrand (WITS) - Vaccines and Infectious Diseases Analytics (VIDA), Johannesburg, Gauteng
  - Wits VIDA Nkanyezi Research Unit, Johannesburg, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Sandton Medical Research Centre, Sandton, Gauteng
  - Gole Biomed Research Centre, Polokwane, Limpopo
  - Merclinco, Middelburg, Mpumalanga
  - Perinatal HIV Research Unit (PHRU), Klerksdorp, North West
  - TREAD Research, Cape Town, Western Cape
  - Tsitsikamma Clinical Research Initiative (TCRI), Plettenberg Bay, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591048